CLINICAL TRIAL: NCT05743374
Title: Micronutrient and Additive Modifications May Optimize Diet To Health
Acronym: Mammoth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Klas Sjöberg, Adjunct professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-01347
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis; Diet Habit; Microbial Colonization
Keywords: Ulcerative colitis; Diet; Microbiota; Emulsifying agent
MeSH Terms: conditions — Colitis, Ulcerative; Feeding Behavior; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Prospective randomized intervention study with elimination of putatively harmful substances in the diet
Who Masked: Participant
Masking Description: Although the patients know that they will be given dietary advice they will not know what type of intervention the other group will be offered. Since dietary advice must be given by the investigators the study cannot be blinded to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal diet (Other): One arm will be given dietary advice that is always given to patients with ulcerative colitis.
  Interventions: Other: Normal diet
- E400 elimination (Active Comparator): The other arm will be given advice to eliminate E400 substances with special regard to carragenan, CMC and polysorbates.
  Interventions: Dietary Supplement: E400 elimination

INTERVENTIONS:
Other: Normal diet — These patients will be given advice about a normal healthy diet.
  Arms: Normal diet
Dietary Supplement: E400 elimination — Patients in the intervention group will be given advice how to eliminate E440 additives with regard to carragenan, CMC and polysorbates.
  Arms: E400 elimination

SUMMARY:
This is a prospective clinical intervention trial where patients with moderately active ulcerative colitis are randomized to either normal healthy diet or a diet with elimination of emulsifying agents within the E 400-group with special respect to carragenan, CMC and polysorbates. At study start and end after one month their diet, clinical characteristics and microbiota will be analysed. The hypotheses are that their disease activity measured with calprotectin and their microbiota will improve after intervention.

DETAILED DESCRIPTION:
Patients with ulcerative colitis attending the out-patient clinic at Skåne university hospital with calprotectin 100-600 will be invited to participate in this diet intervention study. They will be divided into two arms with 35 patients in each, normal diet or E-400 elimination. The diet will be recorded at study start and end with a food diary for four days and a food frequency questionnaire regarding E-400 intake. The patients clinical characteristics (demographics) and disease activity (diarrhoea frequency, blood in stools, abdominal pain, CRP and calprotectin) will be recorded and microbiota collectted. The hypotheses are that the activity measured with clinical characteristics and calprotectin as well as their microboita measured with dysbiosis index and total genom with NGS will improve significantly.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis,
* Moderately active
* Stable medication

Exclusion Criteria:

* Severe disease
* Recent surgery
* Proctitis
* Pregancy
* Treatment with antibiotics
* Difficulties in understanding the information about the study
* Multimorbidity that makes it impossible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2029-06-26 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Calprotectin | One month
  A protein in faeces that increases when there is a flare of the colitis
Microbiota diversity | One month
  The diversity of the GI microbiota reflects disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Klas Sjöberg, Prof, Principal Investigator — Dept of Gastroenterology, SUS, Malmö, Sweden
Locations (1):
- Region Skåne, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
Will be decided based upon cooperation status